CLINICAL TRIAL: NCT06435351
Title: Precision DC: Personalized Neoantigen Dendritic Cell Vaccine Pilot Trial for High Risk Triple Negative Breast Cancer After Neoadjuvant Therapy
Brief Title: Personalized Dendritic Cell Vaccine Pilot for High Risk TNBC After Neoadjuvant Therapy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23142
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Leukapheresis; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dendritic Cell (DC) Vaccine (Experimental): The tumor specimen collected from the primary tumor will undergo whole exome sequencing (WES). The WES data will be analyzed to select up to 20 neoantigens. From this screen up to 10 peptides will be selected to be synthesized for testing and use on the DC pheresis product that will be collected.
  The ready vaccine product will be cryopreserved and then thawed once the patient is ready to under the vaccination sequence.
  Interventions: Procedure: Leukapheresis; Biological: Dendritic Cell (DC) Vaccine

INTERVENTIONS:
Procedure: Leukapheresis — Removal of white blood cells (leukocytes) from the blood. The dendritic cells are harvested from the white blood cells that are collected and trained to recognize the specific abnormal proteins found in the tumor sample.
  One needle is inserted in each arm. An apheresis machine removes blood from the vein in one arm, separates and retains the leukocytes from the blood, and then returns the rest of the blood to the other arm.
Biological: Dendritic Cell (DC) Vaccine — The vaccine will be given intranodally (inguinal or axillary) under ultrasound guidance using a dose of 40-50 million cells three times spaced 2 weeks apart for the initial priming sequence.
  3 doses of the priming vaccines are given once every 2 weeks. 2 booster shots (if available) will be given 6 months and 12 months following completion of initial priming vaccines.

SUMMARY:
This is a pilot protocol to evaluate the safety, feasibility, and immunogenicity of a personalized breast cancer vaccine based utilizing whole exome sequencing data of a patient's residual breast tumor following neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has stage II-III ER/PR less than or equal to 10% HER2 negative by FISH and/or IHC breast cancer treated with standard of care neoadjuvant systemic chemotherapy and surgical resection with significant residual breast tumor (equivalent to RCB II or III) disease.
* Patient has sufficient residual viable primary breast tumor or ipsilateral breast axillary nodal metastatic cancer tissue accessible to Moffitt for whole exome sequencing.
* Patient is 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must have adequate organ and marrow function.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients without radiologic evidence of active metastatic disease and who are within 18 months of their last dose curative intent chemotherapy and/or radiotherapy (whichever is later) for the purposes of study enrollment.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with known active locally advanced unresectable or metastatic cancer.
* Patients with significant uncontrolled intercurrent illness or autoimmune disease requiring systemic immunosuppressants that would be deemed unsuitable to participate in the study by the Principal Investigator (PI).
* Patients who have a medical issue in the opinion of the treating physician and/or PI that would make them unsuitable for pheresis.
* Patients who are currently receiving any other investigational agents.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients enrolled who successfully undergo at least one vaccination. | Up to 3 Years
  Successful production and administration of DC1 priming vaccination sequence in greater than 60% of patients enrolled.

SECONDARY OUTCOMES:
Number of participants who achieve Immunogenicity after administration of vaccine | Up to 3 Years
  Immunogenicity will be determined by ELISpot and reactive T-Cell Receptor (TCR) expansion.
  ELISPot is an enzyme-linked immunospot assay. It is a highly sensitive immunoassay that measures the frequency of cytokine-secreting cells at the single-cell level.
Disease Free Survival (DFS) | Up to 3 Years
  Disease Free Survival will be measured as the length of time after treatment to cancer recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Soliman, MD, Study Director — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/